CLINICAL TRIAL: NCT00762411
Title: Effect of LY450139 a y-Secretase Inhibitor, on the Progression of Alzheimer's Disease as Compared With Placebo
Brief Title: Effects of LY450139, on the Progression of Alzheimer's Disease as Compared With Placebo
Acronym: IDENTITY-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11271; H6L-MC-LFBC (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-01

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — N2-((2S)-2-(3,5-difluorophenyl)-2-hydroxyethanoyl)-N1-((7S)-5-methyl-6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-L-alaninamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LY450139 (Experimental): Participants received 60 milligrams (mg) LY450139 orally once daily for 2 weeks followed by 100 mg LY450139 orally once daily for 2 weeks, then 140 mg LY450139 orally once daily until Week 88.
  Interventions: Drug: LY450139
- Placebo (Placebo Comparator): Participants received placebo orally once daily for the first 76 weeks. At the end of 76 weeks, participants in the placebo arm received LY450139 titrated up to 140 mg orally once daily until Week 88.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY450139 — Administered orally once daily.
  Other Names: Semagacestat
  Arms: LY450139
Drug: Placebo — Administered orally once daily.
  Arms: Placebo

SUMMARY:
Alzheimer's disease (AD) is a fatal degenerative disease of the brain for which there is no cure. AD causes brain cells to die. AD is thought to be caused by an excess of beta amyloid (β-amyloid), a sticky protein in the brain that forms amyloid plaques. At autopsy, AD patients are required to have these amyloid plaques in the brain in order to have a definitive diagnosis of AD. Inhibiting the enzyme gamma-secretase (γ-secretase) lowers the production of β-amyloid. Semagacestat (LY450139) is a functional γ-secretase inhibitor and was shown to lower β-amyloid in blood and spinal fluid in humans tested thus far and in blood, spinal fluid and brain in animals tested thus far. This study used several different tests to measure the effect of semagacestat on both β-amyloid and amyloid plaques for some patients. The buildup of amyloid plaques was measured by a brain scan that takes a picture of amyloid plaques in the brain. Other tests measured the overall function of the brain and brain size in some patients. In this trial, patients who initially received placebo (inactive sugar pill) were, at a certain point in the study, switched over to active drug, semagacestat. In other words, all patients could eventually receive active drug. Each patient's participation could last approximately 2 years. Patients taking approved AD medications were permitted to participate in this study and continue taking these medications during the study. All patients who completed this study had the option to continue receiving semagacestat by participating in an open label study.

Preliminary results from this study (LFBC) (and another similar study LFAN [NCT00594568]) showed semagacestat did not slow disease progression and was associated with worsening of clinical measures of cognition and the ability to perform activities of daily living. Study drug was stopped in all studies. LFBC, LFAN and open label LFBF (NCT01035138) have been amended to continue collecting safety data, including cognitive scores, for at least seven months. The CT-Registry will reflect results of analyses from the original protocol in addition to those from the amended protocol.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for mild to moderate Alzheimer's disease (AD) with Mini-Mental State Examination score of 16 through 26 at visit 1
* Modified Hachinski Ischemia Scale score of less than or equal to 4
* Geriatric Depression Scale score of less than or equal to 6
* A magnetic resonance imaging (MRI) or computerized tomography (CT) scan in the last 2 years with no findings inconsistent with a diagnosis of AD
* If female, must be without menstruation for a least 12 consecutive months or have had both ovaries removed.

Exclusion Criteria:

* Is not capable of swallowing whole oral medication
* Has serious or unstable illnesses
* Does not have a reliable caregiver
* Chronic alcohol and/or drug abuse within the past 5 years
* Has ever had a active vaccination for AD

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1111 (Actual)
Dates: Start 2008-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559 Mon - Fri 9 AM - 5 PM eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (91):
- United States (22):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Costa Mesa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Jolla, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Laguna Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oxnard, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Francisco, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boca Raton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hallandale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hollywood, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Orleans, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shreveport, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hattiesburg, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albany, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manhasset, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
- Brazil (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salvador
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sofia, Bulgaria
- Canada (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint John, New Brunswick
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peterborough, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenfield Park, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Verdun, Quebec
- China (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Xi'an
- France (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poitiers
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
- Germany (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
- Hungary (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Esztergom
- Italy (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boggiovara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cassino
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parma
- Japan (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Akita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Numakunai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aguascalientes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saltillo
- Romania (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Timișoara
- Russia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kazan'
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saratov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yekaterinburg
- Serbia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belgrade
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kragujevac
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon
- Taiwan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changhua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taoyuan District
- Turkey (Türkiye) (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eskişehir
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Istanbul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Izmir
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Samsun
- Ukraine (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dnipropetrovsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Donetsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kherson
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Odesa

REFERENCES:
- [Derived] Liu-Seifert H, Siemers E, Price K, Han B, Selzler KJ, Henley D, Sundell K, Aisen P, Cummings J, Raskin J, Mohs R; Alzheimer's Disease Neuroimaging Initiative. Cognitive Impairment Precedes and Predicts Functional Impairment in Mild Alzheimer's Disease. J Alzheimers Dis. 2015;47(1):205-14. doi: 10.3233/JAD-142508. PMID 26402769
- [Derived] Henley DB, Dowsett SA, Chen YF, Liu-Seifert H, Grill JD, Doody RS, Aisen P, Raman R, Miller DS, Hake AM, Cummings J. Alzheimer's disease progression by geographical region in a clinical trial setting. Alzheimers Res Ther. 2015 Jun 25;7(1):43. doi: 10.1186/s13195-015-0127-0. eCollection 2015. PMID 26120369

RESULTS

PARTICIPANT FLOW:
Groups:
- 140 mg LY450139: Participants received 60 mg LY450139 orally once daily for 2 weeks followed by 100 mg LY450139 orally once daily for 2 weeks, then 140 mg LY450139 orally once daily until Week 88.
Period: Initial Treatment
Arm/Group | 140 mg LY450139 | Placebo
Started | 556 | 555
Intent-to-treat (ITT) | 555 (ITT population included all randomized participants(pts) who received at least 1 dose of study drug.) | 553 (ITT population included all randomized participants who received at least 1 dose of study drug.)
Completed | 22 | 34
Not Completed | 534 | 521
Not completed — Death | 7 | 6
Not completed — Adverse Event | 132 | 40
Not completed — Protocol Violation | 4 | 1
Not completed — Withdrawal by Subject | 65 | 52
Not completed — Physician Decision | 1 | 0
Not completed — Sponsor Decision | 293 | 401
Not completed — Lost to Follow-up | 5 | 0
Not completed — Caregiver Decision | 21 | 16
Not completed — Abnormal Lab/ECG Result | 6 | 4
Not completed — Entry Criteria Exclusion | 0 | 1
Period: Delayed Start
Arm/Group | 140 mg LY450139 | Placebo
Started | 22 | 34
Completed | 5 | 8
Not Completed | 17 | 26
Not completed — Adverse Event | 0 | 4
Not completed — Protocol Violation | 0 | 1
Not completed — Sponsor Decision | 16 | 20
Not completed — Caregiver Decision | 1 | 1
Period: Safety Follow Up (SFU)-Optional
Arm/Group | 140 mg LY450139 | Placebo
Started | 312 (SFU was optional; pts entered from initial treatment and delayed start or did not enter SFU.) | 430 (SFU was optional; pts entered from initial treatment and delayed start or did not enter SFU.)
Completed | 228 | 312
Not Completed | 84 | 118
Not completed — Death | 1 | 8
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 21 | 46
Not completed — Lost to Follow-up | 6 | 1
Not completed — Caregiver Decision | 8 | 8
Not completed — No safety visit or SFU | 48 | 54

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 140 mg LY450139 | Placebo | Total
Number analyzed (Participants) | 555 | 553 | 1108
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.4 (8.0) | 73.0 (8.0) | 73.2 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 316 | 327 | 643
  Male | 239 | 226 | 465
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 358 | 354 | 712
  African | 11 | 8 | 19
  Hispanic | 33 | 29 | 62
  East Asian | 150 | 160 | 310
  West Asian | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  Brazil | 18 | 21 | 39
  Bulgaria | 20 | 18 | 38
  Canada | 50 | 49 | 99
  China | 22 | 22 | 44
  France | 28 | 29 | 57
  Germany | 24 | 20 | 44
  Hungary | 19 | 16 | 35
  Italy | 14 | 11 | 25
  Japan | 64 | 69 | 133
  Korea, Republic of | 38 | 43 | 81
  Mexico | 26 | 24 | 50
  Romania | 20 | 17 | 37
  Russian Federation | 15 | 19 | 34
  Serbia | 5 | 8 | 13
  Taiwan | 25 | 24 | 49
  Turkey | 25 | 23 | 48
  Ukraine | 19 | 20 | 39
  United States | 123 | 120 | 243
Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog11) Score (n=507, 533) [Mean (Standard Deviation); unit: units on a scale] — The cognitive subscale of the ADAS (ADAS-Cog11) consists of 11 items assessing areas of function most typically impaired in AD: orientation, verbal memory, language, and praxis. The scale ranges from 0 to 70, with higher scores indicating greater disease severity.
  units on a scale | 24.5 (9.1) | 24.2 (9.1) | 24.3 (9.1)
Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory Score (n=505, 529) [Mean (Standard Deviation); unit: units on a scale] — The Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL) Inventory Score is a 23-item inventory developed as a rater-administered questionnaire that should be answered by the participant's caregiver. The ADCS-ADL measures both basic and instrumental activities of daily living by participants. The total ADCS-ADL score ranges from 0 to 78, with lower scores indicating greater disease severity.
  units on a scale | 58.8 (13.3) | 59.1 (13.8) | 58.9 (13.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale- Cognitive Subscale (ADAS-Cog11) at 76 Weeks
Description: The cognitive subscale of the ADAS (ADAS Cog11) was used as a primary efficacy measure and consists of 11 items assessing areas of function most typically impaired in Alzheimer's disease (AD): orientation, verbal memory, language, and praxis. The scale ranges from 0 to 70, with higher scores indicating greater disease severity. Least Squares (LS) Mean value was controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (randomization), 76 weeks
Population: Intent to treat (ITT) population: All randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 555 | 553
units on a scale | 7.37 (0.79) | 6.77 (0.72)
Statistical Analysis 1: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.560, Mixed Models Analysis

2. Primary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale- Cognitive Subscale (ADAS-Cog11) at 16 Weeks After Cessation of Study Drug
Description: The cognitive subscale of ADAS (ADAS Cog11) consists of 11 items assessing areas of function most typically impaired in Alzheimer's disease (AD): orientation, verbal memory, language, and praxis. The scale ranges from 0 to 70, with higher scores indicating greater disease severity. Least Squares (LS) Mean value was controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (randomization), 16 weeks following treatment cessation
Population: Intent to treat (ITT) population: All randomized participants who received at least 1 dose of study medication and had both baseline and post-baseline evaluable data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 312 | 430
units on a scale | 4.81 (0.70) | 4.85 (0.63)
Statistical Analysis 1: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.959, Mixed Models Analysis

3. Primary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory (ADCS-ADL) at 76 Weeks
Description: The ADCS-ADL is a 23-item inventory developed as a rater-administered questionnaire answered by the participant's caregiver. The ADCS-ADL measures both basic and instrumental activities of daily living by participants. The total score ranges from 0 to 78, with lower scores indicating greater disease severity. Least Squares (LS) Mean value was controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (randomization), 76 weeks
Population: Intent to treat (ITT) population: All randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 555 | 553
units on a scale | -10.49 (0.98) | -9.77 (0.90)
Statistical Analysis 1: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.567, Mixed Models Analysis

4. Primary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory (ADCS-ADL) at 16 Weeks After Cessation of Study Drug
Description: as for outcome 3
Time Frame: Baseline (randomization), 16 weeks following treatment cessation
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 312 | 430
units on a scale | -8.88 (0.93) | -7.68 (0.84)
Statistical Analysis 1: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.199, Mixed Models Analysis

5. Secondary Outcome: Change From Baseline in Clinical Dementia Rating Sum of Boxes (CDR-SB) at 76 Weeks
Description: CDR-SB is a semi-structured interview of participants and their caregivers. Participant's cognitive status is rated across 6 domains of functioning, including memory, orientation, judgment/problem solving, community affairs, home/hobbies, and personal care. Severity score assigned for each of 6 domains; total score (SB) ranges from 0 to 18. Higher scores indicate greater disease severity. Least Squares (LS) Mean value was controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (randomization), 76 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 22 | 34
units on a scale | 3.05 (1.10) | 4.00 (0.92)
Statistical Analysis 1: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.294, Mixed Models Analysis

6. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) at 76 Weeks
Description: NPI assesses psychopathology in participants with dementia and other neurologic disorders. Information is obtained from a caregiver familiar with the participant's behavior. Total score ranges from 12 to 144; higher scores indicate greater disease severity. Least Squares (LS) Mean value was controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (randomization), 76 weeks
Population: Intent to treat (ITT) population: All randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 555 | 553
units on a scale | 2.94 (1.04) | 3.84 (0.95)
Statistical Analysis 1: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.477, Mixed Models Analysis

7. Secondary Outcome: Change From Baseline in the Resource Utilization in Dementia-Lite (RUD-Lite) up to 76 Weeks
Description: Assesses healthcare resource utilization (formal and informal care). Information gathered on both caregivers (care-giving time, work status) and participants (accommodation and healthcare resource utilization) was gathered from baseline and follow-up interviews. Reported number of hospitalizations per participant up to 76 weeks. Least Squares (LS) Mean value was controlled for age and investigator.
Time Frame: Baseline (randomization), up to 76 weeks
Population: Intent to treat (ITT) population: All randomized participants who received at least 1 dose of study medication, last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: number of hospitalizations
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 555 | 553
number of hospitalizations | 0.72 (0.14) | 0.82 (0.16)
Statistical Analysis 1: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.673, ANCOVA

8. Secondary Outcome: Change From Baseline in the EuroQol 5-Dimensional Health-Related Quality of Life Scale Proxy Version (EQ-5D Proxy) Visual Analog Scale (VAS) at 76 Weeks
Description: EQ-5D (proxy version) measures mobility, self-care, usual activities, pain/discomfort, anxiety/depression; each has 3 severity levels (no, some, severe problems) coded to a 1-digit number (1-3). Digits are combined into 5-digit number describing health state. Numerals 1-3 are not added for total score. VAS assesses caregiver's impression of participant's overall health state; scores range: 0 to 100. Lower scores indicate greater disease severity. Least Squares (LS) Mean value controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (randomization), 76 weeks
Population: Intent to treat (ITT) population: All randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 555 | 553
units on a scale | -4.46 (1.78) | -3.38 (1.64)
Statistical Analysis 1: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.622, Mixed Models Analysis

9. Secondary Outcome: Change From Baseline in Quality of Life in Alzheimer's Disease (QoL-AD) at 76 Weeks
Description: Assess QoL for AD: participant rates mood, relationships, memory, finances, physical condition, and overall QoL assessment. Each of 13 items, rated on a 4-point scale. Sum of items=total score (range: 13 to 52). Higher scores indicate greater QoL. Participant's primary caregiver asked to complete same measure. Least Squares (LS) Mean value controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (randomization), 76 weeks
Population: Intent to treat (ITT) population: All randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 555 | 553
units on a scale | -1.83 (0.47) | -1.05 (0.43)
Statistical Analysis 1: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.178, Mixed Models Analysis

10. Secondary Outcome: Change From Baseline in Mini Mental State Examination (MMSE) at 76 Weeks
Description: MMSE is a brief screening instrument used to assess cognitive function (orientation, memory, attention, ability to name objects, follow verbal/written commands, write a sentence, and copy figures) in elderly participants. Total score ranges from 0 to 30; lower score indicates greater disease severity. Least Squares (LS) Mean value was controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication
Time Frame: Baseline (randomization), 76 weeks
Population: Intent to treat (ITT) population: All randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 555 | 553
units on a scale | -3.56 (0.38) | -3.35 (0.35)
Statistical Analysis 1: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.632, Mixed Models Analysis

11. Secondary Outcome: Percent Change From Baseline in Amyloid Beta (Aβ) 1-42 Plasma Concentration at 52 Weeks
Description: Concentration of amino acid peptide known as Aβ 1-42 in plasma. Least Squares (LS) Mean value was controlled for baseline value, age, and investigator.
Time Frame: Baseline (randomization), 52 weeks
Population: Intent to treat (ITT) population: All randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: picogram per milliliter (pg/mL)
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 555 | 553
picogram per milliliter (pg/mL) | -16.03 (28.33) | 76.37 (24.73)
Statistical Analysis 1: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.009, ANCOVA

12. Secondary Outcome: Change From Baseline in Positron Emission Tomography (PET) Using Fluorine-18 Fluorodeoxyglucose (18F-FDG) at 76 Weeks
Description: Measurement of local cerebral glucose metabolism by PET using the radioactive tracer 18F-FDG. The outcome reported is the composite summary of the standard uptake value ratio (SUVR) normalized to the Pons. Least Squares (LS) Mean value was controlled for baseline value, age, and investigator.
Time Frame: Baseline (randomization), 76 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 74 | 80
ratio | -0.13 (0.05) | -0.08 (0.03)
Statistical Analysis 1: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.426, ANCOVA

13. Secondary Outcome: Change From Baseline in Hippocampal Volume Using Volumetric Magnetic Resonance Imaging (vMRI) up to 76 Weeks
Description: The vMRI assessment of right and left hippocampal volume is reported. Least Squares (LS) Mean value was controlled for baseline value, age, and investigator.
Time Frame: Baseline (randomization), up to 76 weeks
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: cubic millimeter (mm^3)
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 555 | 553
cubic millimeter (mm^3)
  Right Hippocampal Volume | -158.50 (29.44) | -73.60 (24.18)
  Left Hippocampal Volume | -84.41 (61.96) | -111.27 (49.22)
Statistical Analysis 1: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.101, ANCOVA — This is the p-value for the Right Hippocampal Volume
Statistical Analysis 2: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.772, ANCOVA — This is the p-value for the Left Hippocampal Volume

14. Secondary Outcome: Change From Baseline in Amyloid Imaging Positron Emission Tomography (AV-45 PET) up to 76 Weeks
Description: A radioactive tracer for PET that is a ligand for amyloid called [18F]-AV-45. This permits the visualization of amyloid in the brains of Alzheimer's participants. The outcome reported is the composite summary of the standard uptake value ratio (SUVR) normalized to the cerebellar gray matter. Least Squares (LS) Mean value was controlled for baseline value, age, and investigator.
Time Frame: Baseline (randomization), up to 76 weeks
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 555 | 553
ratio | -0.36 (0.23) | 0.16 (0.11)
Statistical Analysis 1: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.326, ANCOVA

15. Secondary Outcome: Change From Baseline in Tau Concentration in Spinal Fluid up to 76 Weeks
Description: Concentration of total tau in spinal fluid. Least Squares (LS) Mean value was controlled for baseline value, age, and investigator.
Time Frame: Baseline (randomization), up to 76 weeks
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: picogram per milliliter (pg/mL)
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 555 | 553
picogram per milliliter (pg/mL) | -11.60 (39.39) | 117.88 (53.58)
Statistical Analysis 1: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.117, ANCOVA

16. Secondary Outcome: LY450139 Population Pharmacokinetics: Clearance of LY450139
Description: Model estimated apparent oral clearance. Clearance is defined as the volume of plasma which is completely cleared of drug (LY450139) per unit time.
Time Frame: 6 weeks, 12 weeks, and 52 weeks
Population: All participants randomized to LY450139 with sufficient dosing information and concentration data to allow estimation of pharmacokinetic parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour (L/h)
Arm/Group | 140 mg LY450139
Number analyzed (Participants) | 517
liters per hour (L/h) | 18.9 (26.6)

17. Secondary Outcome: LY450139 Population Pharmacokinetics: Volume of Distribution of LY450139
Description: Model-estimated apparent volume of distribution. Volume of distribution is a measure of the extent to which drug distributes in the body.
Time Frame: 6 weeks, 12 weeks, and 52 weeks
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters (L)
Arm/Group | 140 mg LY450139
Number analyzed (Participants) | 517
liters (L) | 66.1 (26.2)

18. Secondary Outcome: Change From Baseline in Clinical Dementia Rating Sum of Boxes (CDR-SB) at 4 Weeks After Cessation of Study Drug
Description: Semi-structured interview. Participant's cognitive status rated across 6 domains of functioning: memory, orientation, judgment/problem solving, community affairs, home/hobbies, personal care. Severity score assigned for each of 6 domains; total score (SB) ranges: 0 to 18. Higher scores=greater disease severity. Least Squares Mean value controlled for baseline value, age, investigator, visit, and concomitant standard of care medication. LY450139 dosing stopped due to evidence of dose-dependent cognitive/functional worsening. Participants followed off-dose for 32 weeks, but CDR-SB not assessed.
Time Frame: Baseline (randomization), 4 weeks following treatment cessation
Population: August 2010: all dosing was stopped after protocol-specified interim review showed dose-dependent cognitive/functional worsening of LY450139-treated participants. Participants were followed off-dose for 32 weeks. No analysis was performed at 4 weeks after cessation of drug since this outcome measure was not assessed during the follow-up period.
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) at 4 Weeks After Cessation of Study Drug
Description: NPI assesses psychopathology in participants with dementia and other neurologic disorders. Information is obtained from a caregiver familiar with participant's behavior. Total score ranges from 12 to 144; higher scores indicate greater disease severity. The Least Squares (LS) Mean value was controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication. All LY450139 dosing stopped due to evidence of dose-dependent cognitive/functional worsening. Participants were followed off-dose for 32 weeks, but NPI was not assessed.
Time Frame: Baseline (randomization), 4 weeks following treatment cessation
Population: as for outcome 18
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Change From Baseline in Resource Utilization in Dementia-Lite (RUD-Lite) at 4 Weeks After Cessation of Study Drug
Description: Assesses healthcare resource utilization (formal and informal care). Information gathered on both care-giving time, work status) and participants (accommodation, healthcare resource utilization) is collected. Reported number of participant hospitalizations. Least Squares (LS) Mean value controlled for age and investigator. All LY450139 dosing was stopped due to evidence of dose-dependent cognitive/functional worsening. Participants were followed off-dose for 32 weeks, but RUD-Lite was not assessed.
Time Frame: Baseline (randomization), 4 weeks following treatment cessation
Population: as for outcome 18
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Change From Baseline in EuroQol 5-Dimensional Health-Related Quality of Life Scale Proxy Version (EQ-5D Proxy) Visual Analog Scale (VAS) at 4 Weeks After Cessation of Study Drug
Description: EQ-5D (proxy version) measures mobility, self-care, usual activities, pain/discomfort, anxiety/depression. 3 severity levels: no, some, severe problems. VAS assesses caregiver's impression of participant's health state; score ranges: 0 to 100. Lower scores=greater disease severity. Least Squares (LS) Mean value controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication. All LY450139 dosing was stopped due to evidence of dose-dependent cognitive/functional worsening. Participants were followed off-dose for 32 weeks, but EQ-5D VAS was not assessed.
Time Frame: Baseline (randomization), 4 weeks following treatment cessation
Population: as for outcome 18
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Change From Baseline in Quality of Life in Alzheimer's Disease (QoL-AD) at 4 Weeks After Cessation of Study Drug
Description: Assess QoL for AD; participant rates mood, relationships, memory, finances, physical condition, and overall QoL assessment. Each of 13 items rated on a 4-point scale. Sum of items=total score (range: 13-52). Higher scores=greater QoL. Participant's primary caregiver asked to complete same measure. Least Squares Mean value controlled for baseline, age, investigator, visit, and concomitant standard of care (SOC) medication. All LY450139 dosing was stopped due to evidence of dose-dependent cognitive/functional worsening. Participants were followed off-dose for 32 weeks, but QoL-AD not assessed.
Time Frame: Baseline (randomization), 4 weeks following treatment cessation
Population: as for outcome 18
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Change From Baseline in Mini Mental State Examination (MMSE) 4 Weeks After Cessation of Study Drug
Description: Used to assess cognitive function (orientation, memory, attention, ability to name objects, follow verbal/written commands, write a sentence, and copy figures) in elderly participants. Total score ranges: 0 to 30. Lower score indicates greater disease severity. Least Squares (LS) Mean value was controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication. All LY450139 dosing was stopped due to evidence of dose-dependent cognitive/functional worsening. Participants were followed off-dose for 32 weeks, but MMSE was not assessed.
Time Frame: Baseline (randomization), 4 weeks following treatment cessation
Population: as for outcome 18
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog12) at 76 Weeks
Description: ADAS-Cog12 is ADAS-Cog11 augmented with delayed free recall measure, resulting in a total score ranging from 0 to 80. Higher scores indicate greater disease severity. Least Squares (LS) Mean value was controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (randomization), 76 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 22 | 34
units on a scale | 10.09 (3.29) | 10.34 (2.67)
Statistical Analysis 1: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.929, Mixed Models Analysis

25. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale (ADAS-Cog14) at 76 Weeks
Description: ADAS-Cog14 is ADAS-Cog11 augmented with delayed free recall, digit cancellation, and maze completion measures. A score of 0 to 10 for delayed free recall and a conversion code of 0 to 5 for digit cancellation and maze completion provide total score ranges for this extended ADAS-Cog14 of 0 to 90. Higher scores indicate greater disease severity. Least Squares (LS) Mean value was controlled for baseline value, age, investigator, visit, and concomitant standard of care (SOC) medication.
Time Frame: Baseline (randomization), 76 weeks
Population: Intent to treat (ITT) population: All randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 555 | 553
units on a scale | 9.23 (0.90) | 8.32 (0.82)
Statistical Analysis 1: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.437, Mixed Models Analysis

26. Secondary Outcome: Change From Baseline in Phosphorylated-Tau (P-tau) Concentration in Spinal Fluid up to 76 Weeks
Description: Concentration of p-tau in spinal fluid. Least Squares (LS) Mean value was controlled for baseline value, age, and investigator.
Time Frame: Baseline (randomization), up to 76 weeks
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: picogram per milliliter (pg/mL)
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 555 | 553
picogram per milliliter (pg/mL) | 7.94 (3.06) | 14.75 (4.68)
Statistical Analysis 1: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.318, ANCOVA

27. Secondary Outcome: Change From Baseline in Amyloid Beta (Aβ) 1-42 Concentration in Spinal Fluid up to 76 Weeks
Description: Concentration of an amino acid peptide known as Aβ 1-42 in spinal fluid. Least Squares (LS) Mean value was controlled for baseline value, age, and investigator.
Time Frame: Baseline (randomization), up to 76 weeks
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: picogram per milliliter (pg/mL)
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 555 | 553
picogram per milliliter (pg/mL) | 19.20 (26.03) | -21.39 (35.35)
Statistical Analysis 1: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.417, ANCOVA

28. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog12) at 16 Weeks After Cessation of Study Drug
Description: as for outcome 24
Time Frame: Baseline (randomization), 16 weeks following treatment cessation
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 312 | 430
units on a scale | 5.33 (0.74) | 5.14 (0.67)
Statistical Analysis 1: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.805, Mixed Models Analysis

29. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale (ADAS-Cog14) at 16 Weeks After Cessation of Study Drug
Description: ADAS-Cog14 is ADAS-Cog11 augmented with delayed free recall, digit cancellation, and maze completion measures. A score of 0 to 10 for delayed free recall and a conversion code of 0 to 5 for digit cancellation and maze completion provide total score ranges for this extended ADAS-Cog14 of 0 to 90. Higher scores indicate greater disease severity. Least Squares (LS) Mean value was controlled for baseline value, age, investigator, visit, concomitant standard of care (SOC) medication.
Time Frame: Baseline (randomization), 16 weeks following treatment cessation
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 140 mg LY450139 | Placebo
Number analyzed (Participants) | 312 | 430
units on a scale | 6.00 (0.82) | 5.89 (0.73)
Statistical Analysis 1: Comparison: 140 mg LY450139 vs Placebo; Test type: Superiority or Other; p = 0.893, Mixed Models Analysis

ADVERSE EVENTS:
Groups:
- Placebo- (Initial Treatment Period [NT]): Participants received placebo orally once daily for the first 76 weeks.
- 140 mg LY450139- NT: Participants received 60 mg LY450139 orally once daily for 2 weeks followed by 100 mg LY450139 orally once daily for 2 weeks, then 140 mg LY450139 orally once daily until Week 76.
- Placebo- (Delayed Start Period [DO]): After Week 76, participants received 60 mg LY450139 orally once daily for 2 weeks followed by 100 mg LY450139 orally once daily for 2 weeks, then 140 mg LY450139 orally once daily until Week 88.
- 140 mg LY450139- DO: After Week 76, participants received 140 mg LY450139 orally once daily until Week 88.
- Placebo-Safety Follow Up Period (SFU): For SFU, study drug had been stopped and period was optional to enter; Participants entered from Placebo initial treatment or delayed start or did not enter SFU.
- 140 mg LY450139 - SFU: For SFU, study drug had been stopped and period was optional to enter; Participants entered from 140 mg LY450139 initial treatment or delayed start or did not enter SFU.
Arm/Group | Placebo- (Initial Treatment Period [NT]) | 140 mg LY450139- NT | Placebo- (Delayed Start Period [DO]) | 140 mg LY450139- DO | Placebo-Safety Follow Up Period (SFU) | 140 mg LY450139 - SFU
Serious Adverse Events (participants affected / at risk) | 60/555 | 92/556 | 7/34 | 1/22 | 22/430 | 20/312
Other Adverse Events (participants affected / at risk) | 130/555 | 258/556 | 6/34 | 0/22 | 0/430 | 0/312
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo- (Initial Treatment Period [NT]) (N=555) | 140 mg LY450139- NT (N=556) | Placebo- (Delayed Start Period [DO]) (N=34) | 140 mg LY450139- DO (N=22) | Placebo-Safety Follow Up Period (SFU) (N=430) | 140 mg LY450139 - SFU (N=312)
Anaemia folate deficiency (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 12 (13) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salmonella sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical observation (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/328 (1) | 0/317 (0) | 0/20 (0) | 0/12 (0) | 0/251 (0) | 0/184 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurilemmoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dementia alzheimer's type (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Guillain-barre syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Thalamus haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral caruncle (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0/227 (0) | 1/239 (1) | 0/14 (0) | 0/10 (0) | 0/179 (0) | 1/128 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Activities of daily living impaired (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis obliterans (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo- (Initial Treatment Period [NT]) (N=555) | 140 mg LY450139- NT (N=556) | Placebo- (Delayed Start Period [DO]) (N=34) | 140 mg LY450139- DO (N=22) | Placebo-Safety Follow Up Period (SFU) (N=430) | 140 mg LY450139 - SFU (N=312)
Diarrhoea (Gastrointestinal disorders) | 33 (42) | 58 (72) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 19 (24) | 49 (53) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 17 (22) | 33 (46) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 22 (24) | 28 (31) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0/227 (0) | 0/239 (0) | 1/14 (1) | 0/10 (0) | 0/179 (0) | 0/128 (0)
Weight decreased (Investigations) | 16 (16) | 42 (42) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 16 (16) | 52 (53) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 15 (15) | 30 (32) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 24 (29) | 40 (45) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hair colour changes (Skin and subcutaneous tissue disorders) | 4 (4) | 53 (53) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 5 (6) | 36 (42) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
All dosing for 4-week post-study drug cessation timeframe outcome measures stopped after protocol-specified interim review showed dose-dependent cognitive/functional worsening for LY450139 participants. No assessments made during 32-week follow up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days